CLINICAL TRIAL: NCT01326364
Title: Prognostic Value of Baseline CT Perfusion Parameters of Pancreatic Cancer for Patients Undergoing Stereotactic Body Radiotherapy or Surgical Resection
Brief Title: Prognostic Value of Baseline Computed Tomography (CT) Perfusion Parameters of Pancreatic Cancer for Patients Undergoing Stereotactic Body Radiotherapy or Surgical Resection
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: PANC0009; SU-03182010-5282 (Other: Stanford University)
Record Dates: First submitted 2010-04-14; First posted 2011-03-30 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; iodixanol; Iohexol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Stereotactic body radiotherapy — Standard of Care
  Other Names: CyberKnife
Drug: Iodixanol — IV, calculated per patient
  Other Names: Visipaque
Drug: Iohexol — IV, Calculated per patient
  Other Names: Omnipaque

SUMMARY:
The purpose of this study is first, to determine whether baseline perfusion characteristics of pancreatic cancer, as characterized by CT perfusion studies, can predict tumor response to treatment by stereotactic body radiotherapy (SBRT). The second goal of this study is to determine whether baseline perfusion characteristics in those patients with resectable pancreatic cancer correlate with immunohistologic markers of angiogenesis such as microvessel density and vascular endothelial growth factor (VEGF) expression.

ELIGIBILITY:
Inclusion Criteria:

1. suspected and/or biopsy-proven pancreatic adenocarcinoma, and
2. referral to Radiology for pre-treatment baseline pancreatic protocol CT.

Exclusion criteria:

1) are absolute contraindications to intravenous iodinated contrast or CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pancreatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Histological markers of tumor angiogenesis (microvessel density, EGF/VEGF expression level) | 1 day
Tumor response to treatment in SBRT patients, based on WHO criteria (No Change/Progressive Disease vs. Partial/Complete Response) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aya Kamaya, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States